CLINICAL TRIAL: NCT06541600
Title: Risk Factors for Adverse Outcomes in Sepsis: a Multi-omics Exploration Based on Clinical Cohort Studies
Brief Title: Risk Factors for Adverse Outcomes in Sepsis
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230823
Record Dates: First submitted 2024-05-06; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: sepsis; Septic cardiomyopathy; KKS
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will adopt a retrospective clinical cohort design and include a certain scale of sepsis patients as research objects to find the risk factors for adverse outcomes in patients with sepsis. Bioinformatics techniques were used to infer potential differential genes corresponding to different risk factors. Finally, through the biobank the investigators established in the past, biological samples of patients with sepsis were extracted and protein expression in the samples was detected to comprehensively analyze biological information at multiple levels.

DETAILED DESCRIPTION:
This study was designed as a retrospective single-center clinical study. By searching sepsis patients on the Tongji Cloud platform, the investigators will collect clinical data of patients diagnosed with sepsis from 2003 to 2023 and conduct statistical analysis. In terms of clinical data, the investigators will record the patient's basic information, medical history, clinical symptoms, laboratory results, etc. The main risk factors for adverse clinical outcomes in patients with sepsis were deduced. Through GEO database (GENE EXPRESSION OMNIBUS), bioinformation technology was used to identify the differential genes corresponding to risk factors. Finally, blood samples from sepsis patients were extracted using the biologic specimen bank built by our department of Critical Care Medicine (ethical approval number, No.TJ-IRB20150318) to verify the differential genes from the protein level.

Study population:

This study will select a certain scale of sepsis patients as the study population in order to study the risk factors of adverse outcomes of sepsis from multiple dimensions. The research population criteria the investigators plan to select are as follows: 1. Patients with confirmed Sepsis: Patients participating in this study must meet the clinical diagnostic criteria for sepsis, which means patients with evidence of infection and SOFA score ≥2, according to the definition of Sepsis-3. 2. Age range: The investigators plan to include adults and seniors, with an age range of 18 years and older. Exclusion criteria: Exclude any patient with a cause that causes immune function abnormalities or affects the study results, such as cancer, congenital immune deficiency, autoimmune disease, etc. In addition, the investigators will exclude patients who have other apparently unrelated infections.

For the selection of research groups, the investigators will follow ethical principles and legal provisions to ensure that the research process and the rights and interests of participants are fully protected. The investigators will conduct the research program after obtaining the approval of the Ethics Committee, and protect their privacy and the confidentiality of personal information during the research process. By selecting the appropriate study population, the investigators hope to comprehensively and deeply explore the risk factors for adverse outcomes of sepsis, provide scientific basis for accurate prediction and individualized management, and ultimately improve the prognosis and survival rate of patients with sepsis.

This study will use a multi-omics approach to comprehensively collect and measure data at multiple levels in order to comprehensively understand the risk factors for adverse outcomes in sepsis. The following is what the investigators intend to collect and measure:

1. Clinical data: The investigators will collect the basic information of the patient, including age, gender, BMI, etc. Clinical features associated with sepsis, such as infection site, pathogen type, infection source, complications, etc., will also be collected. In addition, clinical measures associated with adverse outcomes, such as SOFA score, APACHE II score, blood pressure, heart rate, respiratory rate, etc., are also included to assess patient severity and organ function.
2. Biological samples: Blood samples of sepsis patients are extracted from the biobank established by the Department of Critical Care Medicine (ethical approval number, No.TJ-IRB20150318) for subsequent laboratory testing and measurement. The blood samples will be used for gene sequencing, measurement of inflammatory markers, proteomic analysis, and other key indicators including HIF1A (HIF-1 alpha), S100A12 (S100 Calcium-Binding Protein A12), IL-33 (Interleukin-33), HSPA5 (Heat Shock Protein Family A (Hsp70) Member 5), MMP8 (Matrix Metalloproteinase 8), DSC2 (Desmocollin-2), Bradykinin B1 Receptor (BDKRB1), Bradykinin (BK), iNOS (Inducible Nitric Oxide Synthase), etc.
3. Transcriptomics: The data comes from the GEO database, an open data set on the Internet. Through RNA sequencing technology, the investigators will analyze the gene expression profiles of patients at various time points to understand the changes in transcription levels at different stages and under different circumstances. This will help identify biomarkers associated with adverse outcomes and potential therapeutic targets.

In order to ensure the accuracy and consistency of data, the investigators will follow a strict data collection and measurement operation process, and use standardized measurement tools and laboratory techniques to operate. In addition, data quality is strictly controlled during data collection, and data is encrypted and stored to protect patient privacy and personal information.

Finally, through statistical analysis, the investigators hope to identify and quantify the risk factors for adverse outcomes, and provide a scientific basis for prognostic assessment and treatment decisions of patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old;
* meet the diagnostic criteria for sepsis;
* Duration of hospitalization: lasting more than 24 hours;
* no important comorbidities, such as heart failure, liver and kidney insufficiency, malignant tumor, etc.
* Antibiotic use: The time to start antibiotic treatment should not exceed 48 hours.

Exclusion Criteria:

* less than 18 years old;
* Clinical anti-infective therapy: Start long-term anti-infective therapy within 14 days before the expected time point of infection;
* Duration of hospitalization: less than 24 hours;
* The presence of other important complications, such as heart failure, liver and kidney insufficiency, and malignant tumors;
* The presence of other important complications, such as heart failure, liver and kidney insufficiency, and malignant tumors;
* The presence of other infectious diseases, such as tuberculosis, HIV/AIDS, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis
Sampling Method: Probability Sample
Enrollment: 10313 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Survival | 28 days
  Survival
Cardiac function | 24 hours
  Echocardiography (Ejection Fraction (EF))

CONTACTS AND LOCATIONS:
Overall Officials: QIN Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China